CLINICAL TRIAL: NCT04147754
Title: Efficacités comparées du Bloc Des Muscles érecteurs du Rachis, du Bloc péridural et de la rachianalgésie en Chirurgie Thoracique Majeure.
Brief Title: Erector Spinae Block, Epidural Analgesia and Intrathecal Analgesia in Thoracic Surgery
Acronym: SPIRIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019/97
Record Dates: First submitted 2019-10-24; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Surgery
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epidural anesthesia: At physician discretion (observational study)
  Interventions: Procedure: Epidural anesthesia
- Intrathecal morphine: At physician discretion (observational study)
  Interventions: Procedure: Intrathecal morphine
- Erector spinae block: At physician discretion (observational study)
  Interventions: Procedure: Erector spinae block

INTERVENTIONS:
Procedure: Epidural anesthesia — Preoperative epidural anesthesia at physician discretion
  Groups: Epidural anesthesia
Procedure: Intrathecal morphine — Preoperative intrathecal morphine at physician discretion
  Groups: Intrathecal morphine
Procedure: Erector spinae block — Preoperative erector spinae block at physician discretion
  Groups: Erector spinae block

SUMMARY:
Pulmonary thoracic surgery is often responsible for severe postoperative pain, which is associated with an increase in postoperative morbidity and mortality. Moreover, postoperative thoracic pain has a strong impact on patient rehabilitation and is associated with an increase in hospital stay.

Various analgesic techniques allow effective management of pain in the context of thoracic surgery. Regional anesthesia, particularly, allows a powerful analgesia, and limits the use of opioids and their side effects. Among regional anesthesia techniques, thoracic epidural analgesia has become the gold standard for post-thoracotomy analgesia. However, it induces a sympathetic block that promotes in particular per and postoperative hypotension and acute urinary retentions. Thus, new regional anesthesia techniques have been developed and assessed in thoracic surgery in order to avoid side effects related to epidural analgesia, particularly paravertebral block and erector spinae block, but also intrathecal analgesia. Paravertebral block has shown analgesic efficacy after thoracic surgery, and its interest in reducing the risk of hypotension, acute urinary retention, pruritus and postoperative nausea and vomiting compared with the epidural analgesia. Erector spinae block, recently described and evaluated in this context of thoracic surgery, seems to have the same interests and to be easier to achieve than the paravertebral block, but has been little studied. Finally, intrathecal morphine is frequently used because of an easy and rapid realization, and because it allows an adequate analgesia and the reduction of the duration of stay in intensive care compared to the epidural one. However, despite its frequent use, very few studies have compared intrathecal anesthesia with the epidural and other peri-spinal blocks.

These three types of analgesia, epidural analgesia, intrathecal morphine, and erector spinae block are regional anesthesia methods regularly used for pulmonary surgery in the department of the investigators. All of these techniques have shown their analgesic efficacy, but each seems to have particular respective interests, in terms of achievement, management, or perioperative rehabilitation. The objective of the investigators study is to evaluate the effectiveness of each of its techniques to treat postoperative pain and improve the rehabilitation of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic surgery for pulmonary resection
* Scheduled regional anesthesia: epidural anesthesia, intrathecal morphine or erector spinae block

Exclusion Criteria:

* No epidural anesthesia or no intrathecal morphine or no erector spinae block performed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracic surgery for pulmonary resection in the University Hospital of Angers, in France.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-04 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Pain assessment at H+48 | Day 2 after surgery
  Numerical pain rating scale: 0 (no pain at all) to 10 (worst imaginable pain)

SECONDARY OUTCOMES:
Total consumption of morphine (per and postoperative) | Hour 2, Day 1, Day 2 and Day 3 after surgery.
Length of stay in intensive care unit | Through study completion, an average of 1 year
Length of hospital stay | Through study completion, an average of 1 year
Impact on respiratory function | Day 1, Day 2 and Day 3 after surgery.
  Peak Flow in L/min
Frequency of adverse effects related to morphine Frequency of morphine side effects | Hour 2, Day 1, Day 2 and Day 3 after surgery.
Postoperative pain assessment at other times | Hour 2, Day 1, and Day 3 after surgery.
  Numerical pain rating scale: 0 (no pain at all) to 10 (worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Rineau, MD, Principal Investigator — University Hospital of Angers, France
Locations (1):
- CHU Angers - DEPARTEMENT D'ANESTHESIE REANIMATION, Angers, France